CLINICAL TRIAL: NCT00365209
Title: Phase IIA Trial of Curcumin Among Patients With Prevalent Subclinical Neoplastic Lesions (Aberrant Crypt Foci)
Brief Title: Phase II A Trial of Curcumin Among Patients With Prevalent Subclinical Neoplastic Lesions (Aberrant Crypt Foci)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2013-00449; NCI-2013-00449 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UIC-2005-0617; CDR0000483003; UCIRVINE-2005-4586; UIC HS# 2005-0617; CCUM-HUM00000731; P30CA062203 (NIH); 2005-0617 (Other: Chao Family Comprehensive Cancer Center); UCI04-2-01 (Other: DCP); N01CN35160 (NIH)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2014-03

CONDITIONS: Healthy, no Evidence of Disease; Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Curcumin

ARMS (2):
- 2g (curcumin) (Experimental): Patients receive 2 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Other: laboratory biomarker analysis; Other: pharmacological study; Drug: curcumin
- 4g (curcumin) (Experimental): Patients receive 4 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Other: laboratory biomarker analysis; Other: pharmacological study; Drug: curcumin

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: curcumin — Given orally
  Other Names: C.I. 75300; C.I. Natural Yellow 3; CU; Diferuloylmethane

SUMMARY:
Chemoprevention is the use of certain substances to keep cancer from forming, growing, or coming back. Curcumin is a compound found in plants that may prevent colon cancer from forming. This phase II trial is studying how well curcumin works in preventing colon cancer in smokers with aberrant crypt foci.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine mean percentage change from baseline in prostaglandin E2 (PGE2) within ACF pre and post 30 days of curcumin administration at a specified dose.

SECONDARY OBJECTIVS:

I. To determine mean percentage change from baseline in 5-hydroxy-eicosatetraenoic acid (5-HETE) within ACF pre and post 30 days of curcumin administration at a specified dose.

II. To determine mean percentage change from baseline in PGE2 and 5-HETE within comparison normal mucosa pre and post 30 days of curcumin administration at a specified dose.

III. To quantify corresponding enzyme changes in the cyclooxygenases (COX-1, COX-2,) and lipoxygenase (5-LOX) protein abundance. Semi-quantitative changes in these proteins will be measured by western blotting and correlated with changes in prostaglandins and leukotrienes respectively.

IV. Document changes in total ACF number. V. Determine proliferation by Ki-67 IHC in rectal mucosa pre and post therapy and correlate with changes in ACF number and size.

VI. Determine curcumin concentration in rectal mucosa after 30 days therapy and correlate with PGE2 and 5-HETE changes described above.

VII. Measure glutathione peroxidase (GPx) activity within the colon pre and post therapy as an indirect marker of reduced oxidative stress within the colonic epithelium.

VIII. Ensure safety of all participants during course of study investigation. IX. Determine the curcumin concentration in plasma before and after treatment.

OUTLINE: This is a multicenter, nonrandomized, uncontrolled study.

Patients receive 1 of 2 doses of oral curcumin once daily. Treatment continues for 30 days in the absence of unacceptable toxicity or disease progression.

Blood and tissue biopsies are obtained by sigmoidoscopy or colonoscopy at baseline and at day 30 for correlative biomarker studies. The change in prostaglandin E_2 (PGE_2) is assessed by enzyme immunoassay, 5-hydroxy-eicosatetraenoic acid (5-HETE) by high-performance liquid chromatography, cyclooxygenases (COX-1 and COX-2) and 5-lipoxygenase (5-LOX) by western blotting, Ki-67 by immunohistochemistry, and glutathione peroxidase (GPx) by spectrophotometric assay.

After completion of study therapy, patients are followed at 1 week.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker with > 3 pack-year total smoking history
* Subjects taking NSAIDS or ASA < 10 days month are eligible but must undergo 14 day washout and refrain from use during the study
* Subjects who are:

  * Having a clinically indicated screening/surveillance colonoscopy (e.g. due to risk factors, personal history, or symptoms) OR
  * Not having a colonoscopy but are otherwise eligible. These subjects would undergo a flexible sigmoidoscopy.
* ECOG performance status 0-2 (Karnofsky > 60%)
* No severe organ dysfunction which might increase bleeding risk:

  * Demonstrated by: Normal hematologic status (WBC > 3,000/mm^3, hemoglobin > 10.0 gm/dl, and platelet-count >100,000/mm^3), normal hepatic function (bilirubin < 1.5 mg/dl, transaminases < 1.5x institutional norms), and normal renal function (serum creatinine < 2.0 mg/dl, documented in clinical chart 28 days prior to enrollment
* Healthy current smokers (1 cigarette in previous yr) with > 3-pack year of cigarette smoking and able to provide written informed consent; there are no gender restrictions
* The effects of curcumin on the developing human fetus at the recommended therapeutic dose are unknown; for this reason women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* NSAID or ASA use > 10 days /month; any current glucocorticoid use or omega 3-fatty acid supplement use
* Evidence of the following chronic medical conditions such as:

  * Pregnant or lactating women and/or women who are contemplating pregnancy during the duration of the protocol
  * History of chronic inflammatory bowel disease or prior pelvic irradiation
  * History of peptic ulcer disease (PUD) endoscopically confirmed < 5 yrs from enrollment date
  * Newly diagnosed colorectal cancer or advanced adenoma < 1 yr from enrollment
  * Unspecified history of bleeding or coagulation disorder reported by patient or in medical history
  * Hereditary Colon Cancer syndromes (FAP or HNPCC)
* Participants may not be receiving any other investigational agents
* History of contact dermatitis from turmeric
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because curcumin is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with curcumin, breastfeeding should be discontinued if the mother is treated with curcumin

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Meyskens, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 2-stage study. In Stage1, there are 23 enrolled participants who received 2 g curcumin. In Stage2, there are addictional 21 enrolled participants who received 4 g curcumin.
Groups:
- Curcumin: Stage 1: Particpants receive 2 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  Stage 2: Particpants receive 4 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
  curcumin: Given orally
Period: Stage 1: Receiving 2g Curcumin
Arm/Group | Curcumin
Started | 23
Completed | 21
Not Completed | 2
Period: Stage 2: Receiving 4g Curcumin
Arm/Group | Curcumin
Started | 21
Completed | 19
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Stage 1: 2g curcumin (N = 22 participants due to 1 participant withdrew consent after start of treatment) Stage 2: 4g curcumin (N = 21 participants)
Groups:
- Curcumin: Stage 1: Patients receive 2 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  Stage 2: Patients receive 4 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
  curcumin: Given orally
Arm/Group | Curcumin
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years]
  Stage1 2 g (curcumin) N=22 | 57.1 (5.0)
  Stage2 4 g (curcumin) N=21 | 52.2 (6.8)
Sex/Gender, Customized [Number; unit: participants]
  Stage1 2 g (curcumin): Female | 13
  Stage1 2 g (curcumin): Male | 9
  Stage2 4 g (curcumin): Female | 12
  Stage2 4 g (curcumin): Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Baseline in Prostaglandin E2 (PGE2) Within Aberrant Crypt Foci (ACF)
Description: Baseline prostaglandin E2 (PGE2) values found in rectal aberrant crypt foci (ACF) tissue
Time Frame: Baseline
Population: The analysis is based on participants whose data are evaluable and available. Stage1 2 g curcumin: (N = 21 participants) and Stage2 4 g curcumin: (N = 19 participants)
Measure: Mean (Standard Deviation); unit: µg/g protein
Groups:
- Curcumin: Stage 1: Participants receive 2 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  Stage 2: Participants receive 4 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
  curcumin: Given orally
Arm/Group | Curcumin
Number analyzed (Participants) | 40
µg/g protein
  Stage1 2 g (curcumin) N=21 | 1.1 (1.8)
  Stage2 4 g (curcumin) N=19 | 3.4 (4.8)

2. Secondary Outcome: Baseline in 5-hydroxy-eicosatetraenoic Acid (5-HETE) Within Aberrant Crypt Foci (ACF)
Description: Baseline 5-hydroxy-eicosatetraenoic acid (5-HETE) values found in rectal aberrant crypt foci (ACF) tissue
Time Frame: Baseline
Population: The analysis is based on participants whose data are evaluable and available. Stage1 2 g curcumin: (N = 21 participants), Stage2 4 g curcumin: (N = 19 participants)
Measure: Mean (Standard Deviation); unit: µg/g protein
Arm/Group | Curcumin
Number analyzed (Participants) | 40
µg/g protein
  Stage1 2 g (curcumin) N=21 | 1.4 (0.9)
  Stage2 4 g (curcumin) N=19 | 2.3 (1.6)

3. Secondary Outcome: Post-treatment in 5-hydroxy-eicosatetraenoic Acid (5-HETE) Within Aberrant Crypt Foci (ACF)
Description: Post-treatment 5-hydroxy-eicosatetraenoic acid (5-HETE) values found in rectal aberrant crypt foci (ACF) tissue
Time Frame: At 30 Day
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/g protein
Arm/Group | Curcumin
Number analyzed (Participants) | 40
µg/g protein
  Stage1 2 g (curcumin) N=21 | 1.4 (1.0)
  Stage2 4 g (curcumin) N=19 | 1.9 (0.9)

4. Secondary Outcome: Baseline in Prostaglandin E2 (PGE2) Level in Normal Mucosa
Description: Baseline prostaglandin E2 (PGE2) values found in normal mucosa rectal tissue
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/g protein
Arm/Group | Curcumin
Number analyzed (Participants) | 40
µg/g protein
  Stage1 2 g (curcumin) N=21 | 2.1 (3.2)
  Stage2 4 g (curcumin) N=19 | 2.7 (1.9)

5. Secondary Outcome: Post-treatment in Prostaglandin E2 (PGE2) Level in Normal Mucosa
Description: Post-treatment prostaglandin E2 (PGE2) values found in normal mucosa rectal tissue
Time Frame: At 30 day
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/g protein
Arm/Group | Curcumin
Number analyzed (Participants) | 40
µg/g protein
  Stage1 2 g (curcumin) N=21 | 2.7 (3.7)
  Stage2 4 g (curcumin) N=19 | 2.6 (2.9)

6. Secondary Outcome: Baseline in 5-hydroxy-eicosatetraenoic Acid (5-HETE) Level in Normal Mucosa
Description: Baseline 5-hydroxy-eicosatetraenoic acid (5-HETE) values found in normal mucosa rectal tissue
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/g protein
Arm/Group | Curcumin
Number analyzed (Participants) | 40
µg/g protein
  Stage1 2 g (curcumin) N=21 | 2.3 (1.3)
  Stage2 4 g (curcumin) N=19 | 2.5 (1.5)

7. Secondary Outcome: Post-treatment in 5-hydroxy-eicosatetraenoic Acid (5-HETE) Level in Normal Mucosa
Description: Post-treatment 5-hydroxy-eicosatetraenoic acid (5-HETE) values found in normal mucosa rectal tissue
Time Frame: At 30 day
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/g protein
Arm/Group | Curcumin
Number analyzed (Participants) | 40
µg/g protein
  Stage1 2 g (curcumin) N=21 | 2.4 (1.2)
  Stage2 4 g (curcumin) N=19 | 2.2 (1.6)

8. Secondary Outcome: Change in Cyclooxygenases (COX-1, COX-2), and Lipoxygenase (5-LOX) Protein Abundance
Description: The protein levels for each enzyme will be expressed as an absolute change from baseline and graphed against % change of its enzyme product in the same individual. The degree of correlation between these parameters will be assessed by either Pearson's correlation coefficient or Spearman's rank order correlation coefficient.
Time Frame: Baseline to 30 days
Population: There is not enough tissue for the analysis, so no data is provided.
Arm/Group | Curcumin
Number analyzed (Participants) | 0

9. Secondary Outcome: Changes in Total Aberrant Crypt Foci (ACF) Number
Description: Changes in total aberrant crypt foci (ACF) number = Number of ACF at pre-treatment - Number of ACF at post-treatment
Time Frame: Baseline to 30 days
Population: The analysis is based on participants whose data are evaluable and available. Stage1 2 g curcumin: (N = 22 participants), Stage2 4 g curcumin: (N = 19 participants)
Measure: Median (Full Range); unit: Number of ACF
Arm/Group | Curcumin
Number analyzed (Participants) | 41
Number of ACF
  Stage1 2 g (curcumin) N=22 | 0.0 [-18 to 15]
  Stage2 4 g (curcumin) N=19 | 6.0 [-1 to 14]

10. Secondary Outcome: Proliferation by Ki-67 Immunohistochemical Assay (IHC) in Normal Mucosa - Proximal Third
Time Frame: Baseline
Population: The analysis is based on participants whose data are evaluable and available. Stage1 2 g curcumin: (N = 22 participants), Stage2 4 g curcumin: (N = 17 participants)
Measure: Mean (Standard Deviation); unit: percentage of labeled cells
Arm/Group | Curcumin
Number analyzed (Participants) | 39
percentage of labeled cells
  Stage1 2 g (curcumin) N=22 | 0.5 (0.9)
  Stage2 4 g (curcumin) N=17 | 0.3 (0.6)

11. Primary Outcome: Post-treatment in Prostaglandin E2 (PGE2) Within Aberrant Crypt Foci (ACF)
Description: Post-treatment prostaglandin E2 (PGE2) values found in rectal aberrant crypt foci (ACF) tissue
Time Frame: At 30 day
Population: The analysis is based on participants whose data are evaluable and available. Stage1 2g curcumin: (N = 21 participants), Stage2 4 g curcumin: (N = 19 participants)
Measure: Mean (Standard Deviation); unit: µg/g protein
Arm/Group | Curcumin
Number analyzed (Participants) | 40
µg/g protein
  Stage1 2 g (curcumin) N=21 | 1.6 (1.8)
  Stage2 4 g (curcumin) N=19 | 3.7 (3.2)

12. Secondary Outcome: Proliferation by Ki-67 Immunohistochemical Assay (IHC) in Normal Mucosa - Proximal Third
Time Frame: At 30 day
Population: The analysis is based on participants whose data are evaluable and available. Stage1 2 g crucumin: (N = 22 participants), Stage2 4 g curcumin: (N = 19 participants)
Measure: Mean (Standard Deviation); unit: percentage of labeled cells
Arm/Group | Curcumin
Number analyzed (Participants) | 41
percentage of labeled cells
  Stage1 2 g (curcumin) N=22 | 0.6 (1.4)
  Stage 2 4 g (curcumin) N=19 | 0.3 (0.8)

13. Secondary Outcome: Proliferation by Ki-67 Immunohistochemical Assay (IHC) in Normal Mucosa - Middle Third
Time Frame: Baseline
Population: The analysis is based on participants whose data are evaluable and available. Stage1 2 g curcumin: (N = 22 participants), Stage2 4 g curcumin : (N = 17 participants).
Measure: Mean (Standard Deviation); unit: percentage of labeled cells
Arm/Group | Curcumin
Number analyzed (Participants) | 39
percentage of labeled cells
  Stage1 2 g (curcumin) N=22 | 11.9 (4.2)
  Stage2 4 g (curcumin) N=17 | 12.8 (6.1)

14. Secondary Outcome: Proliferation by Ki-67 Immunohistochemical Assay (IHC) in Normal Mucosa - Middle Third
Time Frame: At 30 day
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of labeled cells
Arm/Group | Curcumin
Number analyzed (Participants) | 41
percentage of labeled cells
  Stage1 2 g (curcumin) N=22 | 11.8 (7.2)
  Stage2 4 g (curcumin) N=19 | 16.4 (10.3)

15. Secondary Outcome: Proliferation by Ki-67 Immunohistochemical Assay (IHC) in Normal Mucosa - Distal Third
Time Frame: Baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of labeled cells
Arm/Group | Curcumin
Number analyzed (Participants) | 39
percentage of labeled cells
  Stage1 2 g (curcumin) N=22 | 25.2 (5.3)
  Stage2 4 g (curcumin) N=17 | 28.7 (9.1)

16. Secondary Outcome: Proliferation by Ki-67 Immunohistochemical Assay (IHC) in Normal Mucosa - Distal Third
Time Frame: At 30 day
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of labeled cells
Arm/Group | Curcumin
Number analyzed (Participants) | 41
percentage of labeled cells
  Stage1 2 g (curcumin) N=22 | 23.5 (8.0)
  Stage2 4 g (curcumin) N=19 | 30.9 (7.7)

17. Secondary Outcome: Baseline Curcumin Concentration in Rectal Mucosa
Description: If detectable in the rectal mucosa, it is predicted that curcumin concentrations and potentially curcumin conjugate concentrations will be associated with reduction in PGE2 and 5-HETE measured from colorectal mucosal biopsies. Pearson correlation coefficients between changes in baseline levels in these 2 parameters and curcumin concentration in rectal mucosa will be calculated. Endpoints may be log transformed as appropriate prior to analysis.
Time Frame: Baseline
Population: Samples from 21 participants in the 2g curcumin arm and 18 participants in the 4g curcumin arm were sent to be assayed. Detectable levels of curcumin in rectal mucosa were found in 1 participant in the 2g arm and none in participants on the 4g arm. Therefore, only 1 sample from the 2g arm and 0 samples from the 4g arm are reported here.
Measure: Mean (Standard Deviation); unit: µg/g protein
Units Other Than Participants: samples with detectable levels
Arm/Group | Curcumin
Number analyzed (Participants) | 1
Number analyzed (samples with detectable levels) | 1
µg/g protein | 4.03

18. Secondary Outcome: Post-treatment Curcumin Concentration in Rectal Mucosa
Description: as for outcome 17
Time Frame: At 30 day
Population: The analysis is based on 39 participants (21 participants from 2g curcmin, and 18 participants from 4 g curcumin). In 2g group, a total of 5 samples with detectable levels were analyzed. In 4g group, a total of 3 samples with detectable levels were analyzed.
Measure: Mean (Standard Deviation); unit: µg/g protein
Units Other Than Participants: samples with detectable levels
Arm/Group | Curcumin
Number analyzed (Participants) | 39
Number analyzed (samples with detectable levels) | 8
µg/g protein
  2 g (curcumin) N=21 subjects, N=5 samples analyzed | 8.2 (2.9)
  4 g (curcumin) N=18 subjects, N=3 samples analyzed | 3.8 (0.6)

19. Secondary Outcome: Baseline Curcumin Plasma Concentrations
Description: Baseline curcumin conjugate concentrations will be measured directly from the subject's plasma and then the change in concentrations after the last dose of study drug will be measured. Concentrations will be measured and statistically evaluated by paired t-test or Wilcoxon matched-pairs signed-ranks test, as appropriate.
Time Frame: Baseline
Population: Samples from 19 participants in the 4g curcumin arm were assayed. Detectable levels of curcumin in plasma were found in 4 participants in the 4g arm; therefore, 4 samples are reported here. Samples from participants in the 2g curcumin arm were not collected due to a delayed decision resulting with protocol modification and resource restrictions.
Measure: Mean (Standard Deviation); unit: µg/mL
Units Other Than Participants: samples with detectable levels
Arm/Group | Curcumin
Number analyzed (Participants) | 19
Number analyzed (samples with detectable levels) | 4
µg/mL | 7.3 (8.1)

20. Secondary Outcome: Post-treatment Curcumin Plasma Concentrations
Description: as for outcome 19
Time Frame: At 30 day
Population: Samples from 19 participants in the 4g curcumin arm were assayed. Detectable levels of curcumin in plasma were found in 2 participants in the 4g arm; therefore, 2 samples are reported here. Samples from participants in the 2g curcumin arm were not collected due to a delayed decision resulting with protocol modification and resource restrictions.
Measure: Mean (Standard Deviation); unit: µg/mL
Units Other Than Participants: samples with detectable levels
Arm/Group | Curcumin
Number analyzed (Participants) | 19
Number analyzed (samples with detectable levels) | 2
µg/mL | 3.8 (1.3)

21. Secondary Outcome: Baseline Curcumin Conjugates Concentration in Rectal Mucosa
Description: as for outcome 17
Time Frame: Baseline
Population: Samples from 21 participants in the 2g curcumin arm and 19 participants in the 4g curcumin arm were sent to be assayed. Detectable levels of curcumin conjugates in rectal mucosa were found in 0 participants in the 2g arm and 1 participant on the 4g arm. Therefore, 0 samples from the 2g arm and 1 sample from the 4g arm are reported here.
Measure: Mean (Standard Deviation); unit: µg/g protein
Units Other Than Participants: samples with detectable levels
Arm/Group | Curcumin
Number analyzed (Participants) | 1
Number analyzed (samples with detectable levels) | 1
µg/g protein | 4.21

22. Secondary Outcome: Post-treatment Curcumin Conjugates Concentration in Rectal Mucosa
Description: as for outcome 17
Time Frame: At 30 day
Population: The analysis is based on 39 participants (21 participants from 2g curcumin group and 18 participatns from 4g curcumin group). In 2g group, a total of 13 samples with detectable levels were analyzed. In 4g group, a total of 12 samples with detectable levels were analyzed.
Measure: Mean (Standard Deviation); unit: µg/g protein
Units Other Than Participants: samples with detectable levels
Arm/Group | Curcumin
Number analyzed (Participants) | 39
Number analyzed (samples with detectable levels) | 25
µg/g protein
  2 g (curcumin) N=21 subjects, N=13 samples | 5.9 (2.6)
  4 g (curcumin) N=18 subjects, N=12 samples | 4.5 (1.7)

23. Secondary Outcome: Baseline Curcumin Conjugates Plasma Concentrations
Description: as for outcome 19
Time Frame: Baseline
Population: Samples from 19 participants in the 4g curcumin arm were assayed. Detectable levels of curcumin in plasma were found in 19 participants in the 4g arm; therefore, 19 samples are reported here. Samples from participants in the 2g curcumin arm were not collected due to a delayed decision resulting with protocol modification and resource restrictions.
Measure: Mean (Standard Deviation); unit: µg/mL
Units Other Than Participants: samples with detectable levels
Arm/Group | Curcumin
Number analyzed (Participants) | 19
Number analyzed (samples with detectable levels) | 19
µg/mL | 15.8 (14.8)

24. Secondary Outcome: Post-treatment Curcumin Conjugates Plasma Concentrations
Description: Post-treatment curcumin conjugate concentrations will be measured directly from the subject's plasma and then the change in concentrations after the last dose of study drug will be measured. Concentrations will be measured and statistically evaluated by paired t-test or Wilcoxon matched-pairs signed-ranks test, as appropriate.
Time Frame: At 30 day
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: µg/mL
Units Other Than Participants: samples with detectable levels
Arm/Group | Curcumin
Number analyzed (Participants) | 19
Number analyzed (samples with detectable levels) | 19
µg/mL | 78.5 (84.3)

25. Secondary Outcome: Number of Participants at Each Adverse Event Grade Level
Time Frame: Baseline to 30 days
Population: These participants completed the study. The data is from the final dataset which was available in 2013 following the publication.
Measure: Number; unit: participants
Arm/Group | Curcumin
Number analyzed (Participants) | 41
participants
  2 g (curcumin) N=22: No AE reported | 10
  2 g (curcumin) N=22: AE with a grade of 1 or 2 | 12
  2 g (curcumin) N=22: AE with a grade of 3 | 0
  4 g (curcumin) N=19: No AE reported | 8
  4 g (curcumin) N=19: AE with a grade of 1 or 2 | 10
  4 g (curcumin) N=19: AE with a grade of 3 | 1

ADVERSE EVENTS:
Time Frame: All adverse events are reported and documented from 43 treated participants from the final 2013 dataset. Participants were followed for the duration of the study, an average of 45 days.
Groups:
- Stage1 2 g Curcumin: Stage 1: Participants receive 2 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
  curcumin: Given orally
- Stage2 4 g Curcumin: Stage 2: Participants receive 4 grams of oral curcumin once daily. Treatment continues for up to 30 days in the absence of unacceptable toxicity or disease progression.
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
  curcumin: Given orally
Arm/Group | Stage1 2 g Curcumin | Stage2 4 g Curcumin
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/21
Other Adverse Events (participants affected / at risk) | 12/22 | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage1 2 g Curcumin (N=22) | Stage2 4 g Curcumin (N=21)
ATYPICAL CHEST PAIN (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage1 2 g Curcumin (N=22) | Stage2 4 g Curcumin (N=21)
YELLOW, SOFTER POO (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL CRAMPING (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1)
BEGINNING OF INFLUENZA (General disorders) | 1 (1) | 0 (0)
BURNING WHEN PEE (Renal and urinary disorders) | 1 (1) | 0 (0)
CALMED MY STOMACH (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLD/SINUSES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CURBED APPETITE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
ELEVATED CREATININE (Investigations) | 1 (1) | 0 (0)
EYE VISION IS BLURRY (Eye disorders) | 0 (0) | 1 (1)
FULLNESS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE AT NIGHT (Nervous system disorders) | 0 (0) | 1 (1)
HELPED BOWEL MOVEMENTS, MORE FREQUENT, LOOSER (Gastrointestinal disorders) | 0 (0) | 1 (1)
IMPROVED, EASIER BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 1 (1)
IMPROVED, SOFTER STOOL (Gastrointestinal disorders) | 0 (0) | 1 (1)
IMPROVED; CURCUMIN HELPED CONSTIPATION; BEFORE GOING EVERY 3-4 DAYS, NOW EVERY 2 DAYS (Gastrointestinal disorders) | 0 (0) | 1 (1)
IMPROVED; CURCUMIN WAS BETTER FOR BOWEL MOVEMENT, SOFTER STOOL (Gastrointestinal disorders) | 0 (0) | 1 (1)
IMPROVED; LESS ACHEY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
IMPROVED; MORE FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 (1) | 0 (0)
IMPROVED; NO LONGER CONSTIPATED, CONSTIPATION BEGAN IN 2006; NOW MORE FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 1 (1)
IMPROVED; NOT TOO MUCH GAS IN THE STOMACH (Gastrointestinal disorders) | 0 (0) | 1 (1)
ITCHING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ITCHING ALL OVER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
LEFT AND RIGHT LEG LOWER EDEMA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LITTLE BLOATED (Gastrointestinal disorders) | 0 (0) | 1 (1)
LITTLE BURNING IN STOMACH (Gastrointestinal disorders) | 0 (0) | 1 (1)
LITTLE GAS (Gastrointestinal disorders) | 1 (1) | 0 (0)
LOSS OF APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
LOWER BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MILD HEART BURN (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NO MORE CONSTIPATION, PILL REALLY HELPED (Gastrointestinal disorders) | 0 (0) | 1 (1)
PEEING A LOT (Renal and urinary disorders) | 0 (0) | 1 (1)
PEPPER TASTE (Nervous system disorders) | 1 (1) | 0 (0)
SIDE HURTS (Gastrointestinal disorders) | 1 (1) | 0 (0)
SLOW URINATION (Renal and urinary disorders) | 1 (1) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
STIFFNESS IN NECK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
STOMACH UPSET AND RELATED PAINS (Gastrointestinal disorders) | 1 (1) | 0 (0)
STRAINED SORE CHEST MUSCLES (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
UNUSUAL DREAM STATE (Psychiatric disorders) | 1 (1) | 0 (0)
VOMITTED AFTER TAKING PILLS (Gastrointestinal disorders) | 1 (1) | 0 (0)
WEIRD DREAMS (Psychiatric disorders) | 1 (1) | 0 (0)
YELLOW STOOL (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less